CLINICAL TRIAL: NCT04281524
Title: A Phase 1b, Multi-center, Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy, Safety, and Pharmacokinetics of CSL312 in the Prevention of Peripherally Inserted Central Catheter (PICC)-Associated Thrombosis in Subjects With Cancer
Brief Title: A Clinical Study to Test the Efficacy and Safety of CSL312 on Catheter-associated Blood Clot Formation in Subjects With Cancer Who Receive Chemotherapy Through a PICC Line
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision non-safety related.
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSL312_1002
Record Dates: First submitted 2020-02-21; First posted 2020-02-24 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: PICC-associated Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CSL312 Cohort 1 (Dose 1) (Experimental): CSL312 administered as IV infusion
  Interventions: Drug: CSL312
- CSL312 Cohort 2 (Dose 2) (Experimental): CSL312 administered as IV infusion
  Interventions: Drug: CSL312
- CSL312 Cohort 3 (Dose 3) (Experimental): CSL312 administered as IV infusion
  Interventions: Drug: CSL312
- CSL312 Cohort 4 (Dose 4) (Experimental): CSL312 administered as IV infusion
  Interventions: Drug: CSL312
- Placebo (Placebo Comparator): Placebo administered as IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CSL312 — CSL312 administered as an IV infusion
  Other Names: Garadacimab
  Arms: CSL312 Cohort 1 (Dose 1); CSL312 Cohort 2 (Dose 2); CSL312 Cohort 3 (Dose 3); CSL312 Cohort 4 (Dose 4)
Drug: Placebo — Solution of 70% 0.9% saline / 30% CSL312 diluent
  Arms: Placebo

SUMMARY:
Peripherally Inserted Central Catheters (PICCs) are commonly used in patients with cancer to administer chemotherapy and supportive care medication. However, PICCs and other medical devices that come into contact with blood increase the risk of blood clots (thrombosis) inside the blood vessels. Conventional blood thinners (anticoagulants) may reduce the risk of thrombosis but they also increase the risk of bleeding. CSL312, a monoclonal antibody that inhibits the activated blood clotting factor 12 (FXIIa) will be assessed for its potential to prevent thrombus formation in subjects with cancer at risk of PICC-associated thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older at the time of providing written informed consent
* Diagnosis of malignancy that requires placement of a PICC within the next 3 weeks for administration of chemotherapy (PICC anticipated to be required for at least 1 month)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 [Oken et al, 1982], and investigator's expectation that performance status will remain 0, 1, or 2 for the duration of the study

Exclusion Criteria:

* Active bleeding or with a current clinically significant coagulopathy (eg, international normalized ratio [INR] > 1.5) or clinically significant risk for bleeding (eg, recent intracranial hemorrhage or bleeding peptic ulcer within the last 4 weeks)
* History of venous thrombosis, myocardial infarction or cerebrovascular event within 3 months, or a prothrombotic disorder (eg, antithrombin III, protein C or S deficiency)
* Life expectancy less than study duration (110 days)
* Platelet count of < 20 × 109/L on the day of dose 1 (Day 1) or within 7 days before first dosing
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2
* Treatment with antiplatelet or anticoagulant medication, including thrombosis prophylaxis, within 10 days prior to insertion of the PICC
* Chemotherapy regimen that would be expected to drop the platelet count to < 20 × 109/L
* Chemotherapy regimen with heparin mixed into IV bags (eg, dalteparin 2500 IU/day)
* Difficult IV access that would prevent infusion of the IP
* In situ central venous catheter (CVC) or PICC in the 3 months before the Screening Visit. The study PICC must be inserted in the contralateral side, which must be PICC / CVC naïve
* Undergoing dialysis or have another inserted intravascular foreign surface device
* Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) ≥ 4 × upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with PICC-associated thrombosis | Up to 29 days after PICC insertion
  PICC-associated thrombosis which can be either:
  1. Asymptomatic PICC associated thrombosis detected by Duplex ultrasound (DUS) or venography at Day 15 or Day 29 after PICC insertion or
  2. Symptomatic PICC associated thrombosis up to Day 29 after PICC insertion, suspected clinically due to symptoms of the upper limb or neck, and objectively confirmed by DUS or venography
Percent of subjects with PICC-associated thrombosis | Up to 29 days after PICC insertion
  PICC-associated thrombosis which can be either:
  1. Asymptomatic PICC associated thrombosis detected by Duplex ultrasound (DUS) or venography at Day 15 or Day 29 after PICC insertion or
  2. Symptomatic PICC associated thrombosis up to Day 29 after PICC insertion, suspected clinically due to symptoms of the upper limb or neck, and objectively confirmed by DUS or venography

SECONDARY OUTCOMES:
Overall percentage of subjects with treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | Up to 110 days after first dose of CSL312
Percent of subjects with related TEAEs | Up to 110 days after first dose of CSL312
Percent of subjects with TEAEs by severity | Up to 110 days after first dose of CSL312
Number of subjects treated with CSL312 with detectable antibodies to CSL312 | Up to 110 days after first dose of CSL312
Percent of subjects treated with CSL312 with detectable antibodies to CSL312 | Up to 110 days after first dose of CSL312
Maximum plasma concentration (Cmax) of CSL312 | Up to 110 days after first dose of CSL312
Area under the concentration-time curve (AUC0-t) of CSL312 | Up to 110 days after first dose of CSL312
Time of maximum plasma concentration (Tmax) of CSL312 | Up to 110 days after first dose of CSL312
Terminal elimination half-life (T1/2) of CSL312 | Up to 110 days after first dose of CSL312
Total systemic clearance (CLtot) of CSL312 | Up to 110 days after first dose of CSL312
Volume of distribution during the elimination phase (Vz) of CSL312 | Up to 110 days after first dose of CSL312
Accumulation Ratio (AR) of CSL312 | Up to 110 days after first dose of CSL312
Number of subjects with thrombosis-associated catheter occlusion | Up to 29 days after first dose of CSL312
Percent of subjects with thrombosis-associated catheter occlusion | Up to 29 days after first dose of CSL312
Number of subjects with PICC removal or replacement | Up to 29 days after first dose of CSL312
Percent of subjects with PICC removal or replacement | Up to 29 days after first dose of CSL312
Number of subjects with central line-associated blood stream infections (CLABSI) | Up to 29 days after first dose of CSL312
Percent of subjects with CLABSI | Up to 29 days after first dose of CSL312

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.